CLINICAL TRIAL: NCT04116970
Title: Prospective Trial to Analyze Endobronchial Ultrasound-Guided Transbronchial Needle-Aspiration (EBUS-TBNA) Samples Obtained With and Without Suction
Brief Title: Endobronchial Ultrasound-Guided Transbronchial Needle-Aspiration With Suction in Obtaining Samples From Patients With Suspected Nodal Metastatic Lung Cancer
Acronym: EBUS-Suction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Peter Kneuertz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-18164; NCI-2018-02965 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-09; First posted 2019-10-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (bronchoscopy with EBUS-TBNA with/without vacuum) (Experimental): Patients undergo bronchoscopy with EBUS-TBUA first without and then with applied vacuum.
  Interventions: Procedure: Bronchoscopy; Procedure: Ultrasound-Guided Transbronchial Needle Aspiration

INTERVENTIONS:
Procedure: Bronchoscopy — Undergo bronchoscopy with EBUS-TBNA
Procedure: Ultrasound-Guided Transbronchial Needle Aspiration — Undergo bronchoscopy with EBUS-TBNA
  Other Names: EBUS-TBNA; Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration

SUMMARY:
This trial studies how well endobronchial ultrasound-guided transbronchial needle-aspiration (EBUS-TBNA) with suction works in obtaining samples from patients with suspected lung cancer that has spread to the nodal. EBUS-TBNA samples obtained with additional suction may help to improve material-amounts and decrease blood contamination in the samples.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if suction applied with a vacuum syringe during EBUS-TBNA sampling helps to obtain more material for molecular analyses.

OUTLINE:

Patients undergo bronchoscopy with EBUS-TBUA first without and then with applied vacuum.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography (CT)-scan finding suspicious for lung cancer with nodal metastases
* Clinically stable to undergo diagnostic workup by bronchoscopy with endobronchial ultrasound

Exclusion Criteria:

* Pregnant female
* Minors
* Prisoners
* Patients with contraindication for EBUS such as non-reversible anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of samples collected via endobronchial ultrasound-guided transbronchial needle-aspiration with suction | Up to 3 years
  The qualitative data will have a set number of variable to follow and will be converted to quantitative data. Data will be analyzed using Microsoft Excel, SAS, or SPSS. After checking the normality of the data, all non-parametric data will be converted to parametric data. Appropriate tests for categorical and continuous data will be used. Categorical variables will be compared using Chi-square or Fisher?s Exact test. Normally distributed variables will be compared using Student-T-test and one way analysis of variance. Non-parametric test will include Mann Whitney U test and Kruskal Wallis test. A two tailed p value of < 0.05 will be considered significant.Sample weight (microgram) and visual blood contamination score (0 = no visible blood, 1 = light red shading, 2 = red shading) of endobronchial needle aspiration biopsies obtained with and without suction.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kneuertz, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04116970/ICF_000.pdf